CLINICAL TRIAL: NCT07185438
Title: Efficacy and Safety of Magnetic Resonance Imaging-guided Repetitive Transcranial Magnetic Stimulation (rTMS) in Adolescents With Depression: A Randomized, Double-Blind, Controlled Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Zhou, professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1stChongqingCQMU___ZXY
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Depression - Major Depressive Disorder

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment design. Participants will be randomly assigned in a 1:1:1 ratio to the experimental target rTMS treatment group, the conventional target rTMS treatment group, or the sham stimulation group. All three groups will utilize the Blackdolphin TMS Robot device (SLD-YXRJ) by Xi'an Solide Brain Modulation Ltd. Co., receiving 20 sessions of rTMS stimulation (10 Hz, 120% RMT) or sham stimulation over 4 weeks (with treatment administered on weekdays), with consistent intervention frequency and procedures. Participants will remain in their assigned group for the entire study duration without any crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental target rTMS treatment group (Experimental): Participants will undergo MRI-guided identification of the voxel in the left dorsolateral prefrontal cortex (DLPFC) that is most negatively correlated with the functional connectivity of the subgenual anterior cingulate cortex (sgACC) as the stimulation site. Repetitive transcranial magnetic stimulation (rTMS) (10 Hz, 120% RMT) will be administered using the Blackdolphin TMS Robot device (model SLD-YXRJ) by Xi'an Solide Brain Modulation Ltd. Co., with 20 sessions over 4 weeks (treatment administered on weekdays).
  Interventions: Device: Experimental target rTMS treatment
- Conventional target rTMS treatment group (Experimental): Participants will receive MRI-guided stimulation at the left DLPFC location. Repetitive transcranial magnetic stimulation (rTMS) (10 Hz, 120% RMT) will be administered using the Blackdolphin TMS Robot device (model SLD-YXRJ) by Xi'an Solide Brain Modulation Ltd. Co., with 20 sessions over 4 weeks (treatment administered on weekdays).
  Interventions: Device: Conventional target rTMS treatment
- Sham stimulation treatment group (Sham Comparator): Participants will receive a sham stimulation treatment designed to simulate the rTMS procedure without generating an effective magnetic field output. The intervention will use a dedicated sham stimulation coil, which is identical in appearance, operation, and stimulation protocol to the experimental group. This coil is designed to maintain the same auditory and tactile sensations as the active stimulation but is equipped with an electromagnetic shielding structure or an internal reverse coil arrangement to effectively prevent magnetic flux from penetrating the skull, ensuring no actual neuromodulatory effects.
  Interventions: Device: Sham stimulation treatment

INTERVENTIONS:
Device: Experimental target rTMS treatment — Participants will undergo MRI-guided identification of the voxel in the left dorsolateral prefrontal cortex (DLPFC) that is most negatively correlated with the functional connectivity of the subgenual anterior cingulate cortex (sgACC) as the stimulation site.
  Arms: Experimental target rTMS treatment group
Device: Conventional target rTMS treatment — participants will receive MRI-guided stimulation at the left DLPFC location.
  Arms: Conventional target rTMS treatment group
Device: Sham stimulation treatment — Participants will receive a sham stimulation treatment designed to simulate the rTMS procedure without generating an effective magnetic field output.
  Arms: Sham stimulation treatment group

SUMMARY:
This study aims to assess the feasibility, safety, acceptability, and preliminary efficacy trends of a Magnetic Resonance Imaging-guided Repetitive Transcranial Magnetic Stimulation (rTMS) intervention for adolescent depression through a pilot clinical trial. The findings will inform the design and optimization of subsequent formal randomized controlled trials, providing essential evidence for their execution.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, controlled pilot trial aimed at evaluating the feasibility, safety, acceptability, and preliminary efficacy trends of Magnetic Resonance Imaging-guided Repetitive Transcranial Magnetic Stimulation (rTMS) for the treatment of adolescent depression.

Adolescents diagnosed with Major Depressive Disorder (MDD) will be randomly assigned in a 1:1:1 ratio to one of three groups: the experimental target rTMS treatment group, the conventional target rTMS treatment group, and the sham stimulation group. All three groups will receive 4 weeks of rTMS stimulation (10 Hz, 120% RMT) or sham stimulation intervention, using the Blackdolphin TMS Robot (SLD-YXRJ) by Xi'an Solide Brain Modulation Ltd. Co., with 20 sessions (administered on weekdays) in total. The intervention frequency and procedure will remain consistent across all groups.

In the experimental target rTMS treatment group, participants will undergo MRI-guided identification of the left dorsolateral prefrontal cortex (DLPFC) region, where the voxel most negatively correlated with the functional connectivity of the subgenual anterior cingulate cortex (sgACC) will serve as the stimulation target. In the conventional target rTMS treatment group, participants will receive MRI-guided stimulation at the left DLPFC location. Participants in the sham stimulation group will receive a placebo treatment, simulating the rTMS procedure without generating an effective magnetic field output.

The primary outcome of the treatment phase is the efficacy rate or the remission rate of depressive symptoms. Secondary outcomes include symptom scales, anxiety symptoms, suicide risk, quality of life, sleep, rumination, and cognition. Safety will be monitored through adverse events, vital signs, laboratory tests, and tolerability assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 - 18
2. Diagnosis of major depressive disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), confirmed through the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime version (K-SADS-PL), currently in a depressive episode
3. Score≥40 on the CDRS-R
4. Stable pharmacological treatment: At least 4 weeks of stable psychiatric medication use prior to enrollment, with continuation of the same psychiatric medication regimen throughout the study.

Exclusion Criteria:

1. Psychiatric comorbidities other than anxiety disorders
2. Depression with psychotic symptoms
3. Young Mania Rating Scale (YMRS) score >13
4. A history of neurological disorders (e.g., epilepsy, brain injury) or severe somatic diseases (e.g., thyroid disorders, lupus, diabetes, pulmonary, hepatic, or renal impairment, major trauma)
5. Patients currently using anticonvulsants or high-dose benzodiazepines
6. A history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), or other neuromodulation treatments
7. A history of alcohol or substance abuse or dependence
8. Women who are pregnant or breastfeeding
9. Current high suicide risk
10. Potential complicating factors related to transcranial magnetic stimulation, such as scalp conditions or perforations that may affect magnetic field delivery
11. Contraindications to MRI

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in CDRS-R (Children's Depression Rating Scale) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  Response rate of depressive symptoms (defined as ≥50% reduction in CDRS-R score) or remission rate of depressive symptoms (defined as CDRS-R score ≤28).

SECONDARY OUTCOMES:
Change in BDI-II (Baker Depression Scale) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  Change in BDI-II (Baker Depression Scale) scores from baseline
Change in SCARED (The Screen for Child Anxiety-Related Emotional Disorders) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  Improvement in anxiety (SCARED minus the scores）
Change in suicide risk from baseline on the C-SSRS (Columbia Suicide Severity Rating Scale) | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  The severity of the suicide risk
Change in PSQI (Pittsburgh Sleep Quality Index) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  Improvement in sleep status (PSQI minus the scores）
Change in PedsQL4.0 (The Pediatric Quality of Life Inventory) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  Improvement of children's quality of life（PedsQL4.0 minus the scores)
Change in CGI-S (Clinical Global Impressions-Severity Scales) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  Improvement in overall clinical impression severity（ 7-point scale, with 1 being normal and 7 being among the most severely damaged）
Change in CGI-I (Clinical Global Impressions-Improvement Scales) scores from baseline | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  Improvement of clinical general Impression scale（ 7-point scale,7 denoting a very significant deterioration）
Change in RSS (Ruminative Responses Scale) | Baseline of treatment period, 1 month; The follow-up period was 1 month, 3 months, 6 months.
  The level of improvement in negative thinking（he higher the total score, the more reflective thinking The more severe it is）

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

REFERENCES:
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Croarkin PE, Elmaadawi AZ, Aaronson ST, Schrodt GR Jr, Holbert RC, Verdoliva S, Heart KL, Demitrack MA, Strawn JR. Left prefrontal transcranial magnetic stimulation for treatment-resistant depression in adolescents: a double-blind, randomized, sham-controlled trial. Neuropsychopharmacology. 2021 Jan;46(2):462-469. doi: 10.1038/s41386-020-00829-y. Epub 2020 Sep 12. PMID 32919400
- [Background] Allen CH, Kluger BM, Buard I. Safety of Transcranial Magnetic Stimulation in Children: A Systematic Review of the Literature. Pediatr Neurol. 2017 Mar;68:3-17. doi: 10.1016/j.pediatrneurol.2016.12.009. Epub 2017 Jan 4. PMID 28216033
- [Background] Sigrist C, Vockel J, MacMaster FP, Farzan F, Croarkin PE, Galletly C, Kaess M, Bender S, Koenig J. Transcranial magnetic stimulation in the treatment of adolescent depression: a systematic review and meta-analysis of aggregated and individual-patient data from uncontrolled studies. Eur Child Adolesc Psychiatry. 2022 Oct;31(10):1501-1525. doi: 10.1007/s00787-022-02021-7. Epub 2022 Jun 24. PMID 35751003
- [Background] Berlim MT, Van den Eynde F, Daskalakis ZJ. Efficacy and acceptability of high frequency repetitive transcranial magnetic stimulation (rTMS) versus electroconvulsive therapy (ECT) for major depression: a systematic review and meta-analysis of randomized trials. Depress Anxiety. 2013 Jul;30(7):614-23. doi: 10.1002/da.22060. Epub 2013 Jan 24. PMID 23349112
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] Hetrick SE, McKenzie JE, Bailey AP, Sharma V, Moller CI, Badcock PB, Cox GR, Merry SN, Meader N. New generation antidepressants for depression in children and adolescents: a network meta-analysis. Cochrane Database Syst Rev. 2021 May 24;5(5):CD013674. doi: 10.1002/14651858.CD013674.pub2. PMID 34029378
- [Background] Brent D, Emslie G, Clarke G, Wagner KD, Asarnow JR, Keller M, Vitiello B, Ritz L, Iyengar S, Abebe K, Birmaher B, Ryan N, Kennard B, Hughes C, DeBar L, McCracken J, Strober M, Suddath R, Spirito A, Leonard H, Melhem N, Porta G, Onorato M, Zelazny J. Switching to another SSRI or to venlafaxine with or without cognitive behavioral therapy for adolescents with SSRI-resistant depression: the TORDIA randomized controlled trial. JAMA. 2008 Feb 27;299(8):901-913. doi: 10.1001/jama.299.8.901. PMID 18314433
- [Background] March J, Silva S, Petrycki S, Curry J, Wells K, Fairbank J, Burns B, Domino M, McNulty S, Vitiello B, Severe J; Treatment for Adolescents With Depression Study (TADS) Team. Fluoxetine, cognitive-behavioral therapy, and their combination for adolescents with depression: Treatment for Adolescents With Depression Study (TADS) randomized controlled trial. JAMA. 2004 Aug 18;292(7):807-20. doi: 10.1001/jama.292.7.807. PMID 15315995